CLINICAL TRIAL: NCT04186156
Title: A Phase II Study of Selective HDAC6 Inhibition With KA2507 in Advanced Biliary Tract Cancer Previously Treated With Standard of Care Chemotherapy (ABC-11)
Brief Title: A Study of Selective HDAC6 Inhibition With KA2507 in Advanced Biliary Tract Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not progressing
Sponsor: Karus Therapeutics Limited (Industry)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC-11
Record Dates: First submitted 2019-07-17; First posted 2019-12-04 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KA2507 (HDAC6 inhibitor) (Experimental): This is a single arm dose escalating study. Patients will be treated with open label KA2507 (HDAC6 inhibitor) capsules.
  Interventions: Drug: KA2507

INTERVENTIONS:
Drug: KA2507 — KA2507, an orally-active new chemical entity, is a potent and selective inhibitor of the HDAC6 enzyme, with potential clinical utility in the treatment of melanoma and other solid tumors. KA2507 has been shown to display potent in vitro activity in a range of cancer cell lines, including melanoma cell lines. KA2507 exerts potent in vivo efficacy in a syngeneic model of B16 melanoma. Here, the combination of the agent's direct tumor growth inhibition and metastasis suppression, coupled with its immunotherapeutic activity - demonstrated by decreased expression of STAT-3 and PD-L1 and increased expression of acetylated tubulin, gp100 and MHC Class I in tumors - have been observed.
  Other Names: HDAC6 Inhibitor; HDAC6i

SUMMARY:
To evaluate the preliminary efficacy of KA2507 (an orally active potent and selective HDAC6 inhibitor) in patients with advanced biliary tract cancer (BTC) previously treated with standard of care chemotherapy.

DETAILED DESCRIPTION:
To evaluate the efficacy of KA2507 (an orally active potent and selective HDAC6 inhibitor) in patients with advanced biliary tract cancer (BTC) previously treated with standard of care chemotherapy.

ABC-11 is an open-label, multi-centre study of HDAC6 inhibition using KA2507 in patients with advanced biliary tract cancer previously treated with standard of care chemotherapy.

This is a single-arm single-stage phase II study designed using A'Hern's methodology.

The primary objective of this study is to assess the preliminary efficacy of KA2507 in patients with advanced BTC previously treated with standard of care chemotherapy

A fixed daily dose of KA2507 (800mg BID) will be administered to all patients based on a phase I study, KTP-003.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Signed informed consent
* Histological or cytological diagnosis of advanced (i.e. metastatic disease, or irresectable locally advanced, or recurrent) biliary tract cancer (to include intra or extra hepatic and gall bladder; ampullary cancer will not be included).
* Patient must have disease amenable to biopsy at baseline and consent to pre-treatment biopsy
* Clear evidence of disease progression following standard of care first line therapy with at least 1 measurable lesion using CT/MRI as defined by RECIST 1.1, OR clear evidence of disease progression based on the emergence of non-measurable disease (e.g. new cytologically confirmed ascites, pleural or pericardial effusion)
* Previous treatment with any line of chemotherapy for advanced disease (e.g. currently gemcitabine/cisplatin) OR radiotherapy
* ECOG performance status grade 0-1
* Adequate biliary drainage, with no evidence of ongoing infection
* Estimated life expectancy > 3 months
* Patients intolerant of first-line standard of care chemotherapy will also be eligible provided there is evidence of disease progression

Exclusion Criteria:

* Unresolved or unstable serious toxic side-effects of prior chemotherapy or radiotherapy, i.e. ≥ grade 2 per CTCAE (common terminology criteria for adverse events, v5.0) except fatigue, alopecia and infertility
* Clinical evidence of cerebral metastases
* History of previous malignancy that could interfere with response evaluation
* Concurrent treatment with other investigational drugs within 4 weeks of initiating treatment
* Inadequate renal, liver, or haematological function defined as any of:

  * eGFR < 45 ml/min/1.73 m2 using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula
  * ALT and/or AST > 5 x ULN
  * Neutropenia (absolute neutrophil count < 1.5 x 109/L)
  * Platelets <100 x 109/L
  * Haemoglobin ≤ 9 g/dL). NB the use of transfusion to achieve desired Hb is acceptable
  * Total bilirubin ≥ 1.5 x ULN (except for patients with known Gilbert's syndrome)
* Known haemoglobinopathy due to HbS or HbC disease, α or β thalassemia, or Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Concomitant use of dapsone
* Untreated severe hypothyroidism
* Significant heart disease defined as any of the following:

  * NYHA grade 3 or 4 symptomatic heart failure
  * Unstable angina or acute myocardial infarction within 3 months
  * cardiac ventricular arrhythmia within 3 months that is not controlled by drug therapy and/or by cardiac ablation
  * QTcF > 470 ms on screening ECG or history of Torsades de pointes
* Any other concurrent severe and/or uncontrolled medical or surgical condition which, in the view of the investigator, could compromise the patient's participation in the study
* Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
* Active infection requiring antibiotics within two weeks prior to treatment
* Males who are unable to or refuse to use barrier contraception during treatment and for 3 months after
* Women who are pregnant, breast-feeding or either unable to or refuse to use effective means of contraception during treatment
* Patients who are unable to swallow capsules and/or have a surgical or anatomical condition that precludes swallowing and absorbing oral medication on an ongoing basis
* Any other condition that would, in the investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients alive and progression free at 4 months | 26 months
  Proportion of patients alive and progression free at 4 months (objective disease progression as per RECIST 1.1)

SECONDARY OUTCOMES:
To evaluate tumour response to KA2507 (response rates and duration of response) | 26 months
  To assess the effect of KA2507 on overall response rate according to RECIST Version 1.1.
To evaluate overall survival | 26 months
  Time to death after study treatment.
To characterise the safety and tolerability profile of KA2507 | 26 months
  Incidence of adverse events (Common Terminology Criteria for Adverse Events [CTCAE] Version 5.0)
To characterise the pharmacokinetic profile of KA2507 in a subset of patients | 26 months
  KA2507 plasma pharmacokinetic parameters in plasma from up to six patients.
To determine the pharmacodynamic response to KA2507 | 26 months
  Evidence of selective HDAC6 target engagement inferred through measurement of acetylated tubulin and acetylated histone in peripheral blood T cells from up to six patients

CONTACTS AND LOCATIONS:
Overall Officials: John Bridgewater, Principal Investigator — Cancer Research UK & UCL Cancer Trials Centre
Locations (1):
- Cancer Research UK and UCL Cancer Trials Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No